CLINICAL TRIAL: NCT03058367
Title: Double-blind, Randomised, Three-armed, Placebo-controlled, Clinical Investigation to Evaluate the Benefit and Tolerability of Two Dosages of IQP-AE-103 in Reducing Body Weight in Overweight and Moderately Obese Subjects
Brief Title: Benefit and Tolerability of IQP-AE-103 in Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/023314
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose IQP-AE-103 (1980mg) (Experimental): 2 capsules IQP-AE-103 by mouth, three times a day after main meals for 12 weeks
  Interventions: Dietary Supplement: IQP-AE-103 (330mg)
- Low dose IQP-AE-103 (990mg) (Experimental): 2 capsules IQP-AE-103 by mouth, three times a day after main meals for 12 weeks
  Interventions: Dietary Supplement: IQP-AE-103 (165mg)
- Placebo (Placebo Comparator): 2 capsules IQP-AE-103 by mouth, three times a day after main meals for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AE-103 (330mg) — High dose capsules
  Arms: High dose IQP-AE-103 (1980mg)
Dietary Supplement: IQP-AE-103 (165mg) — Low dose capsules
  Arms: Low dose IQP-AE-103 (990mg)
Dietary Supplement: Placebo — Placebo identical to verum capsules
  Arms: Placebo

SUMMARY:
This study is to evaluate the benefit and tolerability of two dosages of IQP-AE-103 (990mg and 1980mg daily) in reducing body weight in overweight and moderately obese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Overweight to moderately obese subjects (BMI ≥ 25 and < 35 kg/m2)
3. Expressed desire for weight loss
4. Accustomed to 3 main meals/day
5. Commitment to take IP as recommended
6. Commitment to adhere to diet recommendation during the study
7. Commitment to maintain habitual level of activity/exercise during the study
8. Consistent and stable body weight for 3 months prior to V1
9. Commitment to avoid the use of other weight management products or programs during study
10. Commitment and ability to complete the subject diary and study questionnaires
11. Females of childbearing potential: negative pregnancy testing (beta HCG-test in urine) at V1, agreement to use appropriate contraception methods during the study period
12. Consents to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

1. Known sensitivity to the ingredients of the investigational product or source of ingredients
2. Pregnancy or nursing
3. Smoking cessation within 6 months prior to V1 or during the study (regular smoking during the study at the same level as prior to the study is allowed)
4. Current or history of abuse of drugs, alcohol or medication
5. Clinically relevant excursions of safety laboratory parameter
6. Diabetes mellitus type 1
7. Untreated or unstable diabetes mellitus type 2
8. Untreated or unstable endocrine disorders which may influence body weight (e.g. Cushing's disease, thyroid gland disorders)
9. Stenosis in the gastrointestinal (GI) tract
10. Bariatric surgery in subject´s medical history
11. Abdominal surgery within the last 6 months prior to V1
12. Current use of medications that may affect body weight (eg. antipsychotics, anti-depressants, corticosteroids etc.)
13. Presence of acute or chronic gastrointestinal disease (e.g. inflammatory bowel disease, coeliac disease, pancreatitis)
14. Digestion/absorption disorders in gastrointestinal (GI) tract
15. History of eating disorders such as bulimia, anorexia nervosa within the past 12 months prior to V1
16. Other serious organ or systemic diseases such as cancer within the last 5 years prior to V1
17. Any electronic medical implant
18. Use of any medication that could influence GI functions such as antibiotics within 4 weeks and any laxatives, opioids, glucocorticoids, anticholinergics within last 3 months prior to V1 and during the study, as per investigator judgement
19. Any medication or use of products for the treatment of obesity (e.g. orlistat, other fat binder, carbohydrate/starch blocker, fat burner, satiety products etc.) within last 3 months prior to V1 and during the study
20. Participation in similar studies or weight loss programs within last 4 weeks prior to V1
21. Participation in other studies during the last 4 weeks prior to V1
22. Inability to comply
23. Presence of other factor(s) or medication that should preclude subject participation as per investigator judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight (kg) | 12 weeks
  Difference in mean change of body weight (kg) between the higher dosed verum (1980 mg a day) and placebo group after 12 weeks of intervention in comparison to baseline.

SECONDARY OUTCOMES:
Mean change in body weight (kg) | 2, 4, 8, 12 weeks
  Changes in body weight (kg) after 2, 4, 8, and 12 weeks of intervention, each in comparison to baseline, between the two active and placebo group
Mean change in body weight (%) | 2, 4, 8, 12 weeks
  Changes in body weight (%) after 2, 4, 8, and 12 weeks of intervention, each in comparison to baseline, between the two active and placebo group
Proportion of subject weight loss | 2, 4, 8, 12 weeks
  Proportion of subjects who lost at least 3% and 5% of baseline body weight after 2, 4, 8, and 12 weeks intervention, each in comparison to baseline
Change in waist circumference (cm) | 2, 4, 8, 12 weeks
  Changes in waist circumference after 2, 4, 8, and 12 weeks intervention, each in comparison to baseline
Change in hip circumference (cm) | 2, 4, 8, 12 weeks
  Changes in hip circumference after 2, 4, 8, and 12 weeks intervention, each in comparison to baseline

OTHER OUTCOMES:
Safety parameters (lab parameters, vital signs) | 12 weeks
  Change in safety lab parameters, vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Analyze & Realize, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng LV, Cooper J, De Costa P, Chong PW. Microbiota Composition and Diversity in Weight Loss Population After the Intake of IQP-AE-103 in a Double-Blind, Randomized, Placebo-Controlled Study. Front Nutr. 2022 Apr 28;9:790045. doi: 10.3389/fnut.2022.790045. eCollection 2022. PMID 35571928
- [Derived] Uebelhack R, Bongartz U, Seibt S, Bothe G, Chong PW, De Costa P, Wszelaki N. Double-Blind, Randomized, Three-Armed, Placebo-Controlled, Clinical Investigation to Evaluate the Benefit and Tolerability of Two Dosages of IQP-AE-103 in Reducing Body Weight in Overweight and Moderately Obese Subjects. J Obes. 2019 Feb 3;2019:3412952. doi: 10.1155/2019/3412952. eCollection 2019. PMID 30863632